CLINICAL TRIAL: NCT06830850
Title: A Phase I, Open-label, Multi-Center, Non-Randomized Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of HRS-5041 in Subjects With Metastatic Castration-resistant Prostate Cancer
Brief Title: A Trial of HRS-5041-103 to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of HRS-5041 in Subjects With Metastatic Castration-resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-5041-103
Record Dates: First submitted 2025-02-12; First posted 2025-02-17 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Castration Resistant Prostate Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- : HRS-5041 dose level 1 (Experimental): 240 mg BID
  Interventions: Drug: HRS-5041 Single dose of HRS-5041 orally administered

INTERVENTIONS:
Drug: HRS-5041 Single dose of HRS-5041 orally administered — HRS-5041 Oral dosage (Tablet) Oral dosage administration, 28 days per cycle.

SUMMARY:
To evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of 5041-103 in Subjects with Metastatic Castration-resistant Prostate Cancer.

ELIGIBILITY:
IInclusion Criteria

1. Ability to understand the trial procedures and possible adverse events, voluntarily participate in the trial.
2. Adequate bone marrow and other vital organ functions
3. Adequate liver function tests
4. Metastatic Castration-resistant Prostate Cancer

Exclusion Criteria

1. Plan to receive any other anti-tumor therapy during the study.
2. Receipt of any chemotherapy, targeted therapy, immunotherapy, live/attenuated vaccination, radiotherapy or surgery within 4 weeks prior to the first dosing of this study.
3. Uncontrolled hypertension (systolic blood pressure [SBP] > 150 mmHg and/or diastolic blood pressure [DBP] > 100 mmHg with regular anti-hypertension therapy).
4. Factors that may affect the oral administration of the IP (swallow difficulty, chronic diarrhea, and bowel obstruction, etc.), or active gastrointestinal (GI) disease or other disease which may affect the absorption, distribution, metabolism, or elimination of IP.
5. Known history of drug allergies, specific allergies (such as asthma, urticaria, eczema, etc.).
6. Active heart disease within 6 months prior to the first dosing of this study.
7. Medical history of other malignant tumor within 5 years prior to dosing.
8. Positive hepatitis B virus (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C virus (HCV-Ab), or syphilis or severe infections which need treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events, ECOG PS score, vital signs (pulse rate, respiratory rate, blood pressure, body temperature), ECG, clinical chemistry, hematology, urinalysis and physical examination | Screening up to study completion, an average of 1 year.
  To evaluate the safety and tolerability profile of HRS-5041 in subjects with mCRPC.

SECONDARY OUTCOMES:
Concentration | Screening up to study completion,an average of 1 year.
  Plasma concentrations of HRS-5041 during multiple dosing, directly observed from data
Cmax,ss | From administration to C2, up to 4 months.
  Css, max are steady-state maximum concentrations of HRS-5041during multiple dosing, and are directly observed from data.
Cmin,ss | From administration to C2, up to 4 months.
  Css, min are the steady-state trough concentrations of HRS-5041 during multiple dosing, and are directly observed from data
Objective Response Rate (ORR) | Screening up to study completion, an average of 2 years.
  ORR refers to the proportion of subjects with a complete response (CR) or partial response (PR) based on all soft tissue assessments recorded from the date of first drug administration to either the date of radiographic disease progression (including bone progression and soft tissue progression), death from any cause, or the initiation of a new antitumor therapy, whichever occurs first. For subjects with CR or PR at the first evaluation, the efficacy should be confirmed 4 weeks later or at the next tumor imaging evaluation. The numerator includes subjects with a confirmed CR/PR at least 4 weeks after the initial assessment. The denominator consists of subjects with measurable target lesions at baseline.
Best of Response (DoR) | Screening up to study completion, an average of 2 years.
  Best of Response (DoR) BOR refers to the best response of tumor evaluation, including CR, PR, stable disease (SD), progressive disease (PD), and not evaluable for response (NE).
Disease Control Rate (DCR) | Screening up to study completion, an average of 2 years.
  Disease Control Rate (DCR) DCR refers to the time from the first occurrence of CR or PR to PD or death from any cause, whichever occurs first, in subjects with objective response. For subjects who have a confirmed CR or PR, DoR is calculated as the time from the date of first assessment confirming CR or PR to the date of first recorded radiographic disease progression or death from any cause, whichever occurs first. If the subject does not experience PD or death or is lost to follow-up at the end of study, DoR will be censored at the time of the last tumor evaluation.
rPFS (radiographic progression-free survival | Screening up to study completion, an average of 2 years.
  rPFS refers to the time from the first dose of investigational drug to the first radiographic PD or death from any cause (whichever occurs first) as assessed by the investigator. Radiographic disease progression includes both bone progression (based on PCWG3 criteria) and soft tissue progression (based on RECIST v1.1 criteria), with either type of progression counting as progression.
PSA Response Rate at the end of Week 12 | Screening up to the end of Week 12 , up to 4 months.
  Refers to proportion of subjects with a ≥50% decline in serum PSA levels from baseline (PSA50) at the end of 12 weeks of study treatment.
Proportion of Subjects with PSA50 (≥ 50% decline in serum PSA from baseline) | Screening up to the end of treatment, an average of 1 year.
  Refers to proportion of subjects with a ≥50% decline in serum PSA levels from baseline (PSA50) throughout the study treatment period.
Proportion of Subjects with PSA30 (≥ 30% decline in serum PSA from baseline) | Screening up to the end of treatment, an average of 1 year.
  Refers to proportion of subjects with a ≥30% decline in serum PSA levels from baseline (PSA30) throughout the study treatment period.
Time to PSA Progression | From the date of first drug administration to the date of first PSA progression, an average of 1 year.
  Refers to time from the date of first drug administration to the date of first PSA progression. PSA progression is determined based on PCWG3 criteria.
Overall Survival (OS) | From the date of first drug administration to the date of death from any cause, an average of 2 year.
  OS refers to the time from the date of first drug administration to the date of death from any cause. From the date of first drug administration to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (11):
- Australia (11):
  - GenesisCare North Shore (Oncology), Sydney, New South Wales
  - Sydney Adventist Hospital, Sydney, New South Wales
  - Cancer Research SA, Adelaide, South Australia
  - Southern Oncology Clinical Research Unit, Adelaide, South Australia
  - Icon Cancer Centre South Brisbane, Brisbane
  - John Flynn Private Hospital, Brisbane
  - Eastern Health (Box Hill Hospital), Melbourne
  - Linear Clinical Research Ltd, Perth
  - Macquarie University, Sydney
  - MUPharm Pty Limited trading as Macquarie University Hospital Pharmacy, Sydney
  - Illawarra Shoalhaven Local Health District (Wollongong Hospital), Wollongong